CLINICAL TRIAL: NCT00135772
Title: Nicotine and Cotinine Levels in Smokers With Schizophrenia and Schizoaffective Disorder
Brief Title: Nicotine and Cotinine Levels in Smokers With Schizophrenia and Schizoaffective Disorder - 2
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Jill Williams, UMDNJ-Robert Wood Johnson Medical School
Other Study IDs: NIDA-14009-2; K23-14009-2; DPMC
Record Dates: First submitted 2005-08-23; First posted 2005-08-26 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Schizophrenia and Disorders With Psychotic Features; Tobacco Use Disorder
Keywords: nicotine dependence
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Nicotine dependence is very common among individuals with schizophrenia and schizoaffective disorder. Cotinine is a chemical that is made by the body from nicotine. Measuring levels of nicotine and cotinine is an accurate way to determine how much cigarette smoke enters a person's body. The purpose of this study is to measure nicotine and cotinine levels in smokers with schizophrenia or schizoaffective disorder to determine if such individuals absorb more nicotine per cigarette than smokers without schizophrenia-related disorders.

DETAILED DESCRIPTION:
Schizophrenic individuals have higher urinary cotinine levels compared to non-schizophrenic individuals with a similar smoking history. This suggests that schizophrenic individuals may absorb higher doses of nicotine. The purpose of this study is to determine whether smokers with schizophrenia or schizoaffective disorder have higher serum nicotine and cotinine levels in comparison to smokers without schizophrenic-related disorders.

This observational, case-control study will enroll 150 participants, of which 100 will be smokers with schizophrenic-related disorders and 50 will be smokers without a mental illness. Upon completing baseline assessments, participants will smoke a single cigarette. Approximately two minutes following, 3 to 4 ounces of blood will be analyzed for nicotine and cotinine levels. An expired carbon monoxide reading will also be measured. This measurement correlates with the amount of smoke inhalation. Individual participant studies will be completed in 1 to 2 hour-long sessions.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnostic criteria for nicotine dependence and possibly schizophrenia or schizoaffective disorder
* Stable on current antipsychotic regimen(s) for participants with schizophrenia or schizoaffective disorder

Exclusion Criteria:

* At serious risk of suicide, including recent suicidal behavior or attempt within the thirty days prior to study entry
* Current use of clonidine, bupropion, or any other nicotine products (including nicotine patch, gum, inhaler, lozenge or nasal spray)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-10; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M. Williams, M.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ - Robert Wood Johnson Medical School, Piscataway, New Jersey, United States

REFERENCES:
- [Result] Williams JM, Ziedonis DM, Abanyie F, Steinberg ML, Foulds J, Benowitz NL. Increased nicotine and cotinine levels in smokers with schizophrenia and schizoaffective disorder is not a metabolic effect. Schizophr Res. 2005 Nov 15;79(2-3):323-35. doi: 10.1016/j.schres.2005.04.016. Epub 2005 Jun 14. PMID 15961287
- [Result] Williams JM, Gandhi KK, Steinberg ML, Foulds J, Ziedonis DM, Benowitz NL. Higher nicotine and carbon monoxide levels in menthol cigarette smokers with and without schizophrenia. Nicotine Tob Res. 2007 Aug;9(8):873-81. doi: 10.1080/14622200701484995. PMID 17654300